CLINICAL TRIAL: NCT02822495
Title: Expanded Access Protocol for Providing Tabelecleucel to Patients With Epstein-Barr Virus-Associated Viremia or Malignancies for Whom There Are No Appropriate Alternative Therapies
Brief Title: Expanded Access Protocol for Tabelecleucel for Patients With Epstein-Barr Virus-Associated Viremia or Malignancies
Status: No longer available | Type: Expanded Access
Sponsor: Atara Biotherapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ATA129-EAP-901; EBV-CTL-201 (Other: Atara Biotherapeutics)
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Epstein-Barr Virus (EBV) Infections; Lymphoproliferative Disorders; EBV+ Associated Lymphoma; EBV+ Associated Post-transplant Lymphoproliferative Disease (EBV+ PTLD); Epstein-Barr Viremia; Lymphoma, AIDS-related; Epstein-Barr Virus-associated Lymphoproliferative Disease (EBV+ LPD) With Primary Immunodeficiency (PID); Leiomyosarcoma (LMS); Nasopharyngeal Carcinoma (NPC); Epstein-Barr Virus-associated Lymphoproliferative Disease (EBV+ LPD) With Acquired Immunodeficiency (AID); Solid Organ Transplant Complications; Stem Cell Transplant Complications
Keywords: Epstein-Barr Virus (EBV); Solid Organ Transplant (HCT); Hematopoietic Cell Transplant (SOT); Primary Immunodeficiency (PID); Acquired Immunodeficiency (AID); Epstein-Barr Virus-associated Lymphoma; HIV/AIDS Lymphoma; Rheumatoid Arthritis and Lymphoma; Allogeneic, Off-The-Shelf T-cell Immunotherapy; Tumor Necrosis Factor (TNF)-alpha Inhibitors and Lymphoma; Inflammatory Bowel Disease and Lymphoma; Epstein-Barr Virus-specific Cytotoxic T lymphocyte (EBV-CTL); Epstein-Barr Virus+ associated Nasopharyngeal Carcinoma (EBV+ NPC); Epstein-Barr Virus+ associated Leiomyosarcoma (EBV+ LMS)
MeSH Terms: conditions — Epstein-Barr Virus Infections; Infections; Lymphoproliferative Disorders; Lymphoma, AIDS-Related; Leiomyosarcoma; Nasopharyngeal Carcinoma; Primary Immunodeficiency Diseases; Arthritis, Rheumatoid; Lymphoma; Inflammatory Bowel Diseases

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: tabelecleucel — Tabelecleucel is being investigated as an off-the-shelf, allogeneic T-cell immunotherapy for the treatment of EBV+ malignancies and diseases.
  Other Names: tab-cel®; ATA129; EBV-CTL

SUMMARY:
The primary objective of this protocol is to provide expanded access to tabelecleucel to participants with Epstein-Barr virus-associated diseases and malignancies for whom there are no other appropriate therapeutic options, and who are not eligible to enroll in clinical studies designed to support the development and registration of tabelecleucel.

DETAILED DESCRIPTION:
Participants for whom there are no other appropriate therapeutic options and who are not eligible to enroll in other tabelecleucel clinical studies, may be enrolled in this study. After the screening period, participants will receive intravenous infusions of tabelecleucel (1.6 to 2 × 10^6cells/kg) on Day 1, Day 8, and Day 15 of every 35-day cycle. Clinical assessment of disease response is recommended approximately 15 days after the last dose of tabelecleucel to assess the need for additional treatment. The end of expanded access protocol (EAP) visit should be performed at 30 days after the last dose of tabelecleucel.

ELIGIBILITY:
Inclusion Criteria:

1. Any of the following diagnoses of EBV+ malignancies or disease:

   1. EBV+ PTLD following allogeneic hematopoietic cell transplant (HCT)
   2. EBV+ PTLD following solid organ transplant (SOT)
   3. Persistent EBV viremia and known or suspected immunodeficiency
   4. EBV+ LPD that has developed in the setting of an AID
   5. EBV+ LPD that has developed in the setting of a known or suspected PID
   6. EBV+ LMS
   7. EBV+ NPC
2. The evidence of EBV positivity
3. Relapsed or refractory disease, defined as failure to achieve response (ie, complete response or partial response) or recurrent disease following first line therapy, ie, systemic therapy for EBV-related malignancy or viremia for which there are no appropriate therapies.
4. Not eligible for any other Atara clinical development study
5. For participants developing PTLD following allogeneic HCT for acute leukemia, the underlying acute leukemia must be in morphologic remission
6. Adequate organ function per the following:

   1. Absolute neutrophil count >= 500/μL, with or without cytokine support
   2. Platelet count >= 20,000/μL, with or without transfusion support
7. Participant or participant's representative is willing and able to provide written informed consent

Exclusion Criteria:

1. Current diagnosis of Burkitt's lymphoma, classical Hodgkin's lymphoma, or any T-cell lymphoma
2. Prior treatment with any investigational product within 4 weeks of first treatment with tabelecleucel, or within 5 half-lives from the most recent dose to first treatment with tabelecleucel
3. Ongoing need for methotrexate or extracorporeal photopheresis; steroid doses > 1 mg/kg/day of prednisone (or equivalent)
4. Need for vasopressor or ventilatory support, unless deemed to be caused by the EBV-driven process that tabelecleucel is intended to treat
5. Antithymocyte globulin, alemtuzumab, or similar anti-T-cell antibody therapy, or T-cell immunotherapy (donor lymphocyte infusion, other cytotoxic T lymphocytes [CTLs]) <= 4 weeks prior to first treatment with tabelecleucel
6. Pregnancy
7. Female of childbearing potential or male with a female partner of childbearing potential, either of whom are unwilling to use a highly effective method of contraception

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Mehta, DO, Study Director — Atara Biotherapeutics

REFERENCES:
- [Derived] Nikiforow S, Whangbo JS, Reshef R, Tsai DE, Bunin N, Abu-Arja R, Mahadeo KM, Weng WK, Van Besien K, Loeb D, Nasta SD, Nemecek ER, Zhao W, Sun Y, Galderisi F, Wahlstrom J, Mehta A, Gamelin L, Dinavahi R, Prockop S. Tabelecleucel for EBV+ PTLD after allogeneic HCT or SOT in a multicenter expanded access protocol. Blood Adv. 2024 Jun 25;8(12):3001-3012. doi: 10.1182/bloodadvances.2023011626. PMID 38625984